CLINICAL TRIAL: NCT01488162
Title: Non Interventional Study Aimed to Describe the Management of Relapse or Refractory Chronic Lymphocytic Leukemia (CLL) Patients Retreated by MabThera
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Patients With Relapsing or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25664
Record Dates: First submitted 2011-11-04; First posted 2011-12-08 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, prospective, observational study will describe the management of relapsing or refractory chronic lymphocytic leukemia (CLL) patients. Data will be collected for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of relapsed or refractory chronic lymphocytic leukemia (CLL) with first or second relapse
* Previous treatment with MabThera/Rituxan
* MabThera/Rituxan treatment planned for current relapse

Exclusion Criteria:

* Richter syndrome
* Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing or refractory chronic lymphocytic leukemia (CLL)
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2011-04-04 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Chemotherapy regimens associated with MabThera/Rituxan in management of relapse/refractory CLL: Percentage of patients receiving purine analogues/bendamustine/alkylating agents/other chemotherapy | 2 years

SECONDARY OUTCOMES:
Overall response rate | 2 years
Complete response rate | 2 years
Progression-free survival | 2 years
Time to next treatment | 2 years
Overall survival | 2 years
Safety (incidence of adverse events) | 2 years
Safety (incidence of hematologic adverse events) | 2 years
Safety (incidence of infections) | 2 years
Safety (incidence of secondary malignancies) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (67):
- France (67):
  - Aix-en-Provence
  - Albi
  - Angers
  - Antibes
  - Argenteuil
  - Arras
  - Avignon
  - Bayonne
  - Béziers
  - Blois
  - Bobigny
  - Bordeaux
  - Boulogne
  - Bourg-en-Bresse
  - Brest
  - Caen
  - Carcassonne
  - Castelnau Lez
  - Chalon-sur-Saône
  - Chambéry
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Corbeil-Essonnes
  - Creil
  - Fréjus
  - Grenoble
  - La Source
  - La Tronche
  - Le Mans
  - Libourne
  - Lyon
  - Marseille
  - Mâcon
  - Melun
  - Metz
  - Metz-Tessy
  - Montauban
  - Montpellier
  - Mulhouse
  - Nantes
  - Nice
  - Nîmes
  - Paris
  - Perpignan
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Pontoise
  - Reims
  - Rennes
  - Roubaix
  - Rouen
  - Saint Prient En Jarez
  - Saint-Brieuc
  - Saint-Germain-en-Laye
  - Saint-Herblain
  - Saint-Quentin
  - Salon-de-Provence
  - Salouël
  - Strasbourg
  - Toulon
  - Toulouse
  - Tours
  - Troyes
  - Valence
  - Villejuif